CLINICAL TRIAL: NCT04656158
Title: Comparative Effects of Therapeutic Horticulture and Handiwork on Anterior Cingulate Cortex Activation in People With Chronic Low Back Pain : A Randomized Cross-over Controlled Pilot Study
Brief Title: Therapeutic Effects of Horticulture on Anterior Cingulate Cortex Activation in People With Chronic Low Back Pain
Acronym: HORTICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: APHP191119; 2019-A02988-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chronic pain; therapeutic horticulture; anterior cingulate cortex; subgenual prefrontal cortex
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic horticulture (Experimental): handling (gardening equipment) and gardening task (outdoor and greenhouse tasks)
  Interventions: Other: Physical activity involving exposure to nature: Therapeutic horticulture
- Handiwork (Active Comparator): Handling tasks (materials) and handiwork (manufacturing of piece of wooden furniture)
  Interventions: Other: Physical activity involving exposure to nature: Therapeutic horticulture

INTERVENTIONS:
Other: Physical activity involving exposure to nature: Therapeutic horticulture — 2 sessions of 90 minutes of therapeutic horticulture and 2 sessions of 90 minutes of handiwork

SUMMARY:
Chronic low back leads to a significant socio-economic burden. It is associated with physical and psychosocial deconditioning. Even a short "nature experience" has positive effects on the affective and cognitive factors involved in chronic pain. In the brain, the anterior cingulate cortex plays an important role in both pain and emotions. Exposure to a natural environment may decrease activation of the anterior cingulate cortex.

The main objective of this study is to evaluate the effectiveness of therapeutic horticulture on the decrease of activation of the anterior cingulate cortex in people with chronic low back pain participating in 2 sessions of 90 minutes of therapeutic horticulture and 2 sessions of 90 minutes of handiwork.

The investigators hypothesize that therapeutic horticulture may reduce the activation of the anterior cingulate cortex. The effects of therapeutic horticulture may be mediated through the double exposure to both nature and physical activity.

DETAILED DESCRIPTION:
Non-specific low back pain is the first cause of years lived with a disability in the world. The network of biological, psychological and social contributors to chronic low back pain is complex. Within this network, physical and mental deconditioning are a key point and a privileged therapeutic target of multidisciplinary training programs.

Physical exercise improves pain and function in people with chronic low back pain. Nevertheless, its benefits decrease if it is not practiced regularly. The pleasure doing physical exercises and the possibility of integrating them into daily life are important factors of adherence. Gardening meets well the expectations of the physical treatment of chronic low back pain as it involves exercises aiming to increase spinal flexibility, strength and endurance of spine and lower limbs muscles, proprioception. Gardening is associated with the notion of pleasure and can be practiced in a group thus promoting the social bond. Moreover, therapeutic horticulture is suitable for the long term and can even be practiced in urban environment. Painful sensations are modulated by the affective and emotional state. Within the neuromatrix of pain, the cortex plays an important role in encoding pain and associated emotions. Several studies suggest an impact on several physiological parameters of an "experience of nature", even on a short time. A randomized controlled trial compared in 38 healthy volunteers, the effect of a 90-minute walk in nature (forest) and in urban setting (city), on the activation of the anterior cingulate cortex (specifically its subgenual part) assessed using variation in blood perfusion on MRI, and on rumination, assessed using a self-administered questionnaire. The authors showed that neural activation in the subgenual prefrontal cortex and rumination scores were lower in the group of healthy volunteers exposed to nature. Little is known about the impact of a "nature experience" on chronic low back pain. A non-randomized controlled study has shown that adding 7 sessions of therapeutic horticulture to a standardized pain management program improved health status, anxiety and coping strategies in patients with chronic pain.

By its nature and physical component, therapeutic horticulture could constitute a non-pharmacological accurate intervention in people with chronic low back pain, targeting both the neurobiological and physical aspects of deconditioning syndrome. Therapeutic horticulture was introduced in October 2017 in the multidisciplinary training program dedicated to chronic low back pain in our department. However, its effects have not yet been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults of working-age (18 to 70 years),
* Chronic non-specific low back pain,
* Patient waiting for a short functional restoration program in the rehabilitation department,
* Failure of first-line treatment,
* Up-to-date DTP vaccination,
* Patients able to walk 2 km,
* Health insurance,
* Informed written consent.

Exclusion Criteria:

* Specific low back pain,
* Contraindication to MRI,
* Current stoppage or for more than 3 months during the last year,
* Lack of paid employment,
* Participation in another research on low back pain,
* Inability to fluently speak and/or read French language,
* Free state medical assistance
* People under tutorship or curatorship, and protected adults.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Change in the activity of the anterior cingulate cortex | 3 weeks
  The variation in the activity of the anterior cingulate cortex will be measured by the change in blood perfusion in ml / 100 g tissue / min using MRI.

SECONDARY OUTCOMES:
Variation in the rumination score | 3 weeks
  The variation in the rumination score will be measured by means of the self-administered Rumination-Reflection Questionnaire
Variation in the catastrophizing score | 3 weeks
  The catastrophizing score is a sub-scale of the self-administered Coping strategy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin hospital - Department of Physical and Rehabilitation Medicine,, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roren A, Debacker C, Saghiah M, Bedin C, Fayolle A, Abdoul H, Lefevre-Colau MM, Rannou F, Oppenheim C, Nguyen C. Effects of horticultural therapy versus handiwork on anterior cingulate cortex activity in people with chronic low back pain: A randomized, controlled, cross-over, pilot study. PLoS One. 2024 Dec 17;19(12):e0313920. doi: 10.1371/journal.pone.0313920. eCollection 2024. PMID 39689109